CLINICAL TRIAL: NCT02902757
Title: Very Early Response Monitoring in Patients With Glioblastoma Undergoing Therapy Using FDG PET/CT
Brief Title: FDG PET/CT in Monitoring Very Early Therapy Response in Patients With Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-000409; NCI-2016-00583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-000409 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: FDG; PET/CT very early response (48 hrs)
MeSH Terms: conditions — Glioblastoma | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (FDG PET/CT) (Experimental): Patients undergo standard FDG PET/CT scan 6-8 weeks before start of chemotherapy and one additional FDG PET/CT scan within 48 hours of the start of chemotherapy.
  Interventions: Procedure: Computed Tomography; Radiation: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies fluordeoxyglucose (fludeoxyglucose) F-18 (FDG) positron emission tomography (PET)/computed tomography (CT) in monitoring very early therapy response in patients with glioblastoma. Diagnostic procedures, such as FDG PET/CT, may help measure a patient's response to earlier treatment. Chemotherapy can induce very rapid changes to the tumor's glucose consumption which can be measured with imaging. FDG PET/CT shortly after the start of therapy may help identify very early therapy response in patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess very early response to therapy in glioblastoma patients using 18F-FDG PET/CT.

II. Evaluate very early changes in FDG uptake within 48 hours of start of therapy and correlate them with objective response parameters such as Response Assessment in Neuro-Oncology (RANO) and survival.

OUTLINE:

Patients undergo standard FDG PET/CT scan 6-8 weeks before start of chemotherapy and one additional FDG PET/CT scan within 48 hours of the start of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven high grade glioma
* Intention to start therapy

Exclusion Criteria:

* Severe psychiatric illness
* Inability to give written consent
* Breast feeding / pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Changes in glucose uptake | From baseline up to 48 hours
  Standardized uptake values (SUV) will be calculated for different organs and for regions of tumor. Further, regional target to background count-activity ratios will be established.
Very early changes in tumor glucose uptake predictive for objective treatments response and survival assessed using RANO criteria | One PET/CT 48 hours after start of therapy
  SUV will be calculated for different organs and for regions of tumor. Further, regional target to background count-activity ratios will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States